CLINICAL TRIAL: NCT06088550
Title: Effect of Branched-chain Amino Acid Supplementation and Exercise on Quadriceps Muscle Quantity and Quality in Patients With Cirrhosis as Assessed by Ultrasonography
Brief Title: Effect of Branched-chain Amino Acid Supplementation and Exercise on Muscle Quantity and Quality in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasmia Elgohary, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-173-2019
Record Dates: First submitted 2023-08-26; First posted 2023-10-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Muscle Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group-1 (No Intervention): received standard care
- Group-2 (Active Comparator): received BCAA
  Interventions: Dietary Supplement: BCAA
- Group-3 (Active Comparator): Recieved Exercice
  Interventions: Other: home-based graded exercise program
- Group-4 (Active Comparator): Received a combined BCAA + Exercise
  Interventions: Dietary Supplement: BCAA; Other: home-based graded exercise program

INTERVENTIONS:
Dietary Supplement: BCAA — a branched-chain amino acid (BCAA) formula: taken by oral route in the form of 2 scoops of Protofit BCAA daily on 200 cc water, (manufactured by Dulex lab company). Each scoop contains 5 gm BCAA (2.5 gm leucine, 1.25 gm isoleucine & 1.25 gm valine).
  Arms: Group-2; Group-4
Other: home-based graded exercise program — home-based graded exercise program comprises both aerobic and resistance exercise. The exercise was done by the patients themselves aided by a physiotherapist, a nurse or patients' relatives
  Arms: Group-3; Group-4

SUMMARY:
Introduction: Ultrasound can be used to monitor muscle mass during interventional approaches in patients with liver cirrhosis.

The aim: To investigate the effect of branched-chain amino acid (BCAA) supplementation and/or muscle exercise on ultrasound-measured quadriceps muscle thickness and echo intensity, as well as on muscle strength, performance, and nutritional assessment in patients with cirrhosis.

Patients & Methods: This is a randomized controlled study that included 220 liver cirrhosis patients with Child-Pugh B & C classes. They were randomized into a control group comprising 55 patients who received only the standard care, and interventional groups comprising 165 patients equally distributed into three groups, they received in addition to standard care, BCAA, programmed exercise, or BCAA and programmed exercise respectively. At baseline and after 28 days, all participants were subjected to ultrasound-measured quadriceps muscle thickness and echo intensity, in addition to handgrip strength, short physical performance battery (SPPB), anthropometric measures, hematological and biochemical assessment, MELD score measurement, nutritional assessment using 7- subjective global assessment score (SGA).

DETAILED DESCRIPTION:
This is an open, 4-arm parallel, randomized controlled trial conducted on cirrhotic patients

All eligible patients received instructions of standard care that includes standard diet and non-exercise activity thermogenesis (NEAT), then the patients were randomly assigned in an allocation ratio of approximately 1:1:1:1; group 1= control received the standard care only, and three intervention groups; group 2 received added 10 gm/day branched-chain amino acid (BCAA) (manufactured by Dulex lab company). Group 3 received added home-based exercise comprising both aerobic and resistance exercises, and finally, group 4 received added both BCAA and home-based exercise.

All patients were subjected to the following at the baseline and after 28 days:

1. thorough medical history
2. Complete clinical examination including BP, middle upper arm circumference (MUC), and body mass index (BMI) using the dry weight.
3. The nutritional status assessment using the 7-point Subjective Global Assessment (SGA) score,
4. Assessment of their physical fitness using the short physical performance battery test (SPPB) score.
5. Assessment of muscle strength using handgrip strength using a digital dynamometer (Model: 12-0286).
6. Routine labs including complete blood count (CBC), liver function, kidney function, and electrolytes, FBG
7. Calculation of Child-Pugh & MELD scores.
8. Ultrasound assessment of quadriceps muscle thickness and echogenicity

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with moderate and marked liver impairment

Exclusion Criteria:

* cirrhotic patients with Child-Pugh class A, patients with acute liver cell failure or malignancies, associated other end-organ failure, and vitally unstable patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
a change from baseline of muscle quantity | 28 days
  assessed by ultrasound quadriceps muscle thickness
a change from baseline of muscle strength | 28 days
  assessed by handgrip strength
a change from baseline of muscle performance | 28 days
  assessed by the short physical performance battery test (SPPB)
a change from baseline of muscle quality | 28 days
  assessed by ultrasound quadriceps muscle echo intensity

SECONDARY OUTCOMES:
a change from the baseline of nutritional status | 28 days
  assessed by 7-point Subjective Global Assessment (SGA) score
a change from the baseline of MELD score | 28 days
  assessed by calculating MELD score at baseline and after 28 days
a change from the baseline of ascites | 28 days
  assessed by subjective clinical grading
a change from the baseline of hematological parameters | 28 days
  assessed by CBC
a change from the baseline of liver enzymes | 28 days
  assessed by laboratory assessment of liver enzymes
a change from the baseline of BP | 28 days
  assessed by measuring BP
a change from the baseline edema | 28 days
  assessed by clinical grading

CONTACTS AND LOCATIONS:
Overall Officials: Elham Sobhy, Principal Investigator — Kasr Alainy School of Medicine
Locations (1):
- Kasr Aliny School of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sobhy E, Kamal MM, Saad Y, Saleh DA, Elgohary R, Hassan MS. Effect of branched-chain amino acid supplementation and exercise on quadriceps muscle quantity and quality in patients with cirrhosis as assessed by ultrasonography: A randomized controlled trial. Clin Nutr ESPEN. 2024 Jun;61:108-118. doi: 10.1016/j.clnesp.2024.03.011. Epub 2024 Mar 15. PMID 38777422